CLINICAL TRIAL: NCT01546883
Title: Dabigatran-related Effect on Progression of Atrial Fibrosis in Patients With Atrial Fibrillation
Brief Title: Dabigatran's Effect on Changes in Atrial Fibrosis in Patients With Atrial Fibrillation
Acronym: DEPAF
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Not enough patients in time period allotted for study
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Nassir F. Marrouche, MD, Associate Professor, University of Utah
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: IRB # 43119
Record Dates: First submitted 2012-02-15; First posted 2012-03-07 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Atrial Fibrillation
Keywords: Atrial fibrillation; MRI
MeSH Terms: conditions — Atrial Fibrillation | interventions — Dabigatran

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Dabigatran (Experimental): Patients with Atrial fibrillation taking Dabigatran etexilate as the anti-coagulant
  Interventions: Drug: Dabigatran etexilate (Pradaxa)

INTERVENTIONS:
Drug: Dabigatran etexilate (Pradaxa) — 150mg bid or 75mg bid for a period of one year
  Other Names: Pradaxa

SUMMARY:
This study includes treating patients with atrial fibrillation (AF) with Dabigatran, an anti-coagulant for a period of one year to see if there are any significant changes in the degree of left atrial structural remodeling in these patients. The investigators hypothesize that there will be a significant decrease in the degree of left atrial structural remodeling (fibrosis) in AF patients treated with dabigatran.

DETAILED DESCRIPTION:
Atrial fibrillation (AF) is one of the most common cardiac arrhythmia in medical practice in both the clinical and hospital settings. In addition to a three-fold increase in the risk of mortality, AF patients are at an increased risk of developing a stroke. This risk increased from 6.7% for those who are 50-59 years of age to 36.2% for those between 80-89 years of age. One of the most serious complications of AF is thromboembolism (TE), including both Transient Ischemic Attack (TIA) and stroke, which can be fatal or disabling in many patients and is associated with either type of AF - recurrent or persistent. Image-based methods of risk-stratification and clinical scoring systems, such as the CHADS2 score, have the potential to advance our understanding of the mechanisms governing AF recurrence as well as thrombus formation and can improve our ability to prevent these potentially devastating complications.

Treatments for AF include antiarrhythmic drug therapy, anticoagulation, catheter ablation, and cardioversion, all of which have been thoroughly studied. Anticoagulation is undisputably effective in preventing strokes in patients with AF, reducing the incidence of stroke by 3 fold in high-risk patients. Pradaxa® (Dabigatran etexilate) is a new oral anticoagulant that was approved by the FDA on October 19, 2010 for reducing the risk of stroke and systemic embolism in patients with non-valvular AF. Pradaxa is a direct and reversible inhibitor of thrombin, the penultimate protease in the coagulation process. Thrombin converts fibrinogen to fibrin, which participates in forming the matrix of blood clots. Pradaxa® inhibits formation of thrombus by inhibiting the conversion of fibrinogen to fibrin. Prior to approval of Pradaxa®, warfarin has been the only other oral anticoagulant available in the US for reducing the risk of stroke associated with AF, but its use is limited because of a number of undesirable characteristics. Recently, the RE-LY study showed Pradaxa® 150mg bid was statistically significantly superior to warfarin in reducing the risk of strokes in patients with AF, although there was no statistically significant difference in risk of hemorrhage between warfarin and Pradaxa®. Pradaxa® will be used for its approved indication in this study.

The link between AF and stroke is complex but remodeling of the left atrium (LA) may play a central role. Atrial remodeling refers to any persistent change in atrial structure and function. Fibrosis, an extensive deposition of extracellular matrix components (specifically collagen and fibronectin), is the major causative component of structural remodeling of LA. AF promotes fibrosis and this structural remodeling in turn leads to increased heterogeneity of electrical conduction in the LA which can contribute to AF progression. Late gadolinium enhancement magnetic resonance imaging (LGE-MRI), is a noninvasive technique that allows us to detect and quantify structural remodeling of the LA tissue in patients with AF . Changes in the composition of LA tissue is detected by LGE-MRI based on the delayed enhancement property of the gadolinium-based contrast agent, whose slow washout kinetics relative to normal surrounding tissue, can be quantified as increased fibrosis (structural remodeling of myocardium prior to any ablation) or scar (inflammation and tissue remodeling post ablation). Preliminary findings from our lab demonstrate a significantly larger amount of atrial remodeling / fibrosis detected using LGE-MRI in those patients with strokes compared to those without.

Thrombin (the protease inhibited by Pradaxa®), also is a potent mitogen for connective-tissue producing cells which are prone to developing fibrosis and a chemoattractant for fibroblasts, thus playing an important role in development of tissue fibrosis. Bogatkevich et al. recently demonstrated Pradaxa restrained fibrotic events in lung fibroblasts, suggesting that thrombin inhibition could be an effective strategy for inhibiting fibrosis in other organs, including the heart.

We suggest the characteristics of the fibrosis that we quantify in the left atrium will be similar to the fibrosis seen in the other organs such as lungs, skin and kidney. We hypothesize that Pradaxa will inhibit left atrial structural remodeling (measured as percent fibrosis) associated with AF.

In this study, we plan to study the effect of Pradaxa on remodeling of left atrial structure (measured as percent fibrosis) as detected by LGE-MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with all types of non-valvular AF (includes paroxysmal, persistent and permanent AF)
2. Candidate for anticoagulation therapy
3. No contra-indication for LGE-MRI
4. Patients age 18 and older
5. Patients who are able to provide informed consent to participate in the study

Exclusion Criteria:

1. Patients who have already undergone an atrial fibrillation ablation procedure.
2. Patients with active contra-indications to any anticoagulant agent.
3. Other major bleeding disorders or risk factors that would place the patient at risk of bleeding.
4. Recent surgery (within 30 days).
5. Renal insufficiency, severe kidney disorders/diseases, GFR < 30mg/dL (Gadolinium contraindication).
6. Advanced liver disease.
7. Any health related Gadolinium/MRI contraindications: Pacemaker devices, etc.
8. Pregnant, planning to be become pregnant or nursing women
9. Individuals who are unable to provide informed consent
10. Contraindicated for Pradaxa® .
11. Patients the Investigators feel are inappropriate for the study
12. Patients who cannot give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2012-02; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nassir F Marrouche, MD, FHRS, Principal Investigator — University of Utah, CARMA center
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: medical clinic
Period: Overall Study
Arm/Group | Dabigatran
Started | 14
Completed | 2
Not Completed | 12
Not completed — Withdrawal by Subject | 3
Not completed — Adverse Event | 4
Not completed — Lost to Follow-up | 2
Not completed — early closure of study | 2
Not completed — other unrelated illness | 1

BASELINE CHARACTERISTICS:
Groups:
- Dabigatran: Dabigatran
Arm/Group | Dabigatran
Number analyzed (Participants) | 14
Age, Continuous [Mean (Standard Deviation); unit: years] | 60 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10
  Male | 4
Region of Enrollment [Number; unit: participants]
  United States | 14

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Fibrosis
Description: We will measure the change in percentage of fibrosis over a one-year period when drug is taken. We will calculate the results as percentage of fibrosis measured using MRI at 12 months minus the percentage of fibrosis measured using MRI at baseline to clarify if there is a decrease in fibrosis in the one year period.
Time Frame: MRI at baseline and MRI at 12 months post-enrollment
Population: Data were not collected for the analysis population and therefore could not be summarized to include in this report.
Arm/Group | Dabigatran
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Groups:
- Dabigatran: Patients taking Dabigatran
Arm/Group | Dabigatran
Serious Adverse Events (participants affected / at risk) | 1/14
Other Adverse Events (participants affected / at risk) | 9/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran (N=14)
GI bleed (Gastrointestinal disorders) | 1 (1) — Patient suffered a GI bleed which was later determined to be expected and not associated with the study.
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Dabigatran (N=14)
abdominal pain (Gastrointestinal disorders) | 2 (2)
respiratory tract infection (Infections and infestations) | 1 (1)
urinary tract infection (Infections and infestations) | 1 (1)
rectal bleeding (Gastrointestinal disorders) | 1 (1)
lesions on tongue (Gastrointestinal disorders) | 1 (1)
shortness of breath, dizziness, fatigue (General disorders) | 3 (3)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days